CLINICAL TRIAL: NCT04021121
Title: Pharmacokinetics and Tolerability of Adjunctive Linezolid for the Treatment of Tuberculous Meningitis
Brief Title: Adjunctive Linezolid for the Treatment of Tuberculous Meningitis
Acronym: ALTER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: MRC/UVRI and LSHTM Uganda Research Unit (Other); London School of Hygiene and Tropical Medicine (Other); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 18-26068; R21TW011035 (NIH)
Record Dates: First submitted 2019-06-03; First posted 2019-07-16 (Actual); Results first posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Tuberculosis, Meningeal
MeSH Terms: conditions — Tuberculosis, Meningeal | interventions — Linezolid; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- High Dose RIF with LZD (Experimental): Arm 1 participants will receive high dose oral RIF (35mg/kg/day) and LZD 1200 mg daily for the first 4 weeks of therapy, along with standard doses of Isoniazid (INH), Pyrazinamide (PZA), and Ethambutol (EMB). After 4 weeks, LZD will be discontinued and high dose RIF will return to standard dose for the remainder of treatment.
  Interventions: Drug: LZD; Drug: High dose RIF
- Standard dose RIF with LZD (Experimental): Arm 2 participants will receive standard dose RIF, INH, PZA, and EMB along with LZD 1200 mg daily. After 4 weeks, LZD will be discontinued.
  Interventions: Drug: LZD; Drug: Standard dose RIF
- High Dose RIF (Experimental): Arm 3 participants will receive high dose oral RIF (35mg/kg/day) for the first 4 weeks of therapy, along with standard doses of INH, PZA, and EMB. After 4 weeks, high dose RIF will return to standard dose for the remainder of treatment.
  Interventions: Drug: High dose RIF
- Standard Dose RIF (Active Comparator): Arm 4 participants will receive standard doses of RIF, INH, PZA, and EMB.
  Interventions: Drug: Standard dose RIF

INTERVENTIONS:
Drug: LZD — LZD 1200 mg daily
  Other Names: Linezolid
  Arms: High Dose RIF with LZD; Standard dose RIF with LZD
Drug: High dose RIF — RIF 35 mg/kg/day
  Arms: High Dose RIF; High Dose RIF with LZD
Drug: Standard dose RIF — RIF 10 mg/kg/day
  Arms: Standard Dose RIF; Standard dose RIF with LZD

SUMMARY:
This is a phase II randomized open-label trial of high versus standard dose rifampin (RIF) with or without linezolid (LZD) for the first 4 weeks of treatment for Tuberculosis Meningitis (TBM) at Masaka Regional Referral Hospital in Uganda. Initial randomization will be to high (35 mg/kg/day) versus standard (10 mg/kg/day) dose oral rifampin for the first 4 weeks of intensive therapy. Participants will then undergo a second randomization to linezolid 1200 mg daily versus no linezolid for the first 4 weeks of therapy. The primary aims are (1) to determine the cerebrospinal fluid and plasma pharmacokinetics of adjunctive LZD 1200 mg daily in TBM patients receiving high or standard dose RIF and (2) to evaluate the tolerability of a 4-week course of LZD in TBM patients.

ELIGIBILITY:
Inclusion Criteria

1. Age > 18 years
2. Written informed consent from participant or proxy
3. Definite, probable, possible, or suspected TBM diagnosis wherein the patient is being committed to a full course of anti-TB treatment for TBM in the setting of routine care.

All participants must have at least one of the following signs/symptoms: headache, irritability, vomiting, fever, neck stiffness, convulsions, focal neurological deficits, altered consciousness, or lethargy. In addition, participants must have CSF glucose to plasma ratio < 0.5 OR positive CSF acid-fast bacilli (AFB) smear OR positive CSF GeneXpert or Xpert Ultra OR clinician intent to initiate TB treatment for suspected TB meningitis.

Definite, probable and possible TBM will be defined as:

Definite TBM is defined by the presence of one or more of the following:

* Acid- fast bacilli (AFB) seen in the CSF, M tuberculosis cultured from CSF, or a CSF M tuberculosis-positive nucleic acid amplification test (e.g., Gene Xpert Ultra) performed within 14 days of entry
* AFB seen in the context of histological changes consistent with tuberculosis in the brain with suggestive symptoms or signs and CSF changes.

Probable and possible TBM are defined using previously published consensus criteria as shown in Appendix A45.

* Probable TBM is defined as a total score of ≥12 when neuroimaging is available or total score of ≥10 when neuroimaging is unavailable. At least two points should either come from CSF or cerebral imaging criteria.
* Possible TBM is defined as a total score of 6-11 when neuroimaging is available, or total score of 6-9 when neuroimaging is unavailable.

Exclusion of the most likely alternative diagnoses is also required (e.g., negative cryptococcal antigen). Because culture confirmation is rarely available or often delayed in TBM, patients with probable or possible TBM will be recruited based on these predefined criteria, and CSF will be collected for mycobacterial culture and molecular testing. Classification of participants as definite, probable, or possible TBM will be made retrospectively once all necessary data are available.

Exclusion criteria

1. >5 doses of TB treatment received within previous 5 days
2. Discontinued TB treatment in prior 14 days
3. Known current/previous drug resistant TB infection
4. Known allergy to RIF, INH, PZA, EMB, LZD
5. Previous treatment of TB or TBM with LZD
6. Concomitant or planned use of monoamine oxidase inhibitors, selective serotonin reuptake inhibitors, HIV protease inhibitors, or any other drug with significant interaction with RIF, LZD, or any TB drugs (see Appendices C and D)
7. Women who are pregnant or breastfeeding, or women or men of reproductive potential who are unwilling to use at least one reliable form of barrier contraception or to abstain from sexual activity while receiving study drug treatment and for 30 days after stopping study treatment. Acceptable forms of contraception include: condoms (male or female) with or without a spermicidal agent, or diaphragm or cervical cap with spermicide. Hormonal contraception is not recommended as it may be ineffective due to induction of metabolism when receiving rifampicin.
8. Unwillingness to be an inpatient for 2 weeks for initial treatment or to attend follow up clinic visits
9. Lack of informed consent from participant or next of kin/caregiver
10. Serum creatinine >1.8 times upper limit of normal, hemoglobin <7.0 g/dL for men, <6.5 g/dL for women, platelet count <50,000/mm3, absolute neutrophil count <600/mm3, alanine aminotransferase (ALT) >3 times the upper limit of normal, total bilirubin >2 times the upper limit of normal.
11. Severe peripheral neuropathy defined by Grade 3 symptoms AND vibratory loss OR absent ankle jerks for participants able to undergo the Brief Peripheral Neuropathy Screen (see Appendix B).
12. Contraindication to LP, including PLT <50 cells/mm3 or unequal pressures between intracranial compartments (e.g., due to mass lesion, non-communicating hydrocephalus), or unwillingness to undergo or consent to LP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Felicia C Chow, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Masaka Regional Referral Hospital/MRC UVRI Uganda Research Unit on AIDS, Masaka, Uganda

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High Dose RIF With LZD | Standard Dose RIF With LZD | High Dose RIF | Standard Dose RIF
Started | 9 | 11 | 10 | 10
Completed | 6 | 8 | 5 | 6
Not Completed | 3 | 3 | 5 | 4
Not completed — Death | 3 | 3 | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose RIF With LZD | Standard Dose RIF With LZD | High Dose RIF | Standard Dose RIF | Total
Number analyzed (Participants) | 9 | 11 | 10 | 10 | 40
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 39 [36 to 42] | 35 [33 to 43] | 38 [28 to 42] | 33 [27 to 42] | 37 [29 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 8 | 6 | 6 | 22
  Male | 7 | 3 | 4 | 4 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 9 | 11 | 10 | 10 | 40
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Living with HIV infection [Count of Participants; unit: Participants] | 9 | 11 | 9 | 10 | 39

OUTCOME MEASURES:

1. Primary Outcome: Drug Clearance (CL/F)
Description: Parameters were estimated in NONMEM v7.5 using maximum likelihood estimation (MLE) by optimizing the likelihood function based on observed data. The First Order Conditional Estimation (FOCE) method was employed, which linearizes the model around individual-specific estimates to efficiently account for both fixed effects (population-level parameters) and random effects (individual variability).
Time Frame: 4 weeks
Population: Our primary outcomes include only 2 out of the 4 arms (High dose RIF with LZD + Standard Dose with LZD) because only these 2 arms received linezolid (LZD), and the primary outcomes are measures of LZD pharmacokinetics. Thus, the other 2 arms (High dose RIF with No LZD + Standard Dose with No LZD) are not relevant. Additionally, as pre-specified in the protocol, the 2 arms that received LZD (High dose RIF with LZD + Standard Dose with LZD) are combined.
Measure: Mean (95% Confidence Interval); unit: L/hr
Groups:
- Linezolid: Includes arm 1 (Linezolid, high dose rifampicin) and arm 2 (Linezolid, standard dose rifampicin)
Arm/Group | Linezolid
Number analyzed (Participants) | 18
L/hr | 6.24 [5.305 to 7.175]

2. Primary Outcome: Volume of Distribution (Vd)
Description: as for outcome 1
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: L
Arm/Group | Linezolid
Number analyzed (Participants) | 18
L | 24.97 [14.024 to 35.976]

3. Primary Outcome: Plasma Absorption Rate Constant (ka)
Description: as for outcome 1
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: per hour (hr^-1)
Arm/Group | Linezolid
Number analyzed (Participants) | 18
per hour (hr^-1) | 0.35 [.173 to .527]

4. Primary Outcome: Rate of CSF Uptake (kPC)
Description: as for outcome 1
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: per hour (hr^-1)
Arm/Group | Linezolid
Number analyzed (Participants) | 18
per hour (hr^-1) | 0.382 [.278 to .486]

5. Primary Outcome: CSF to Plasma Ratio (PC)
Description: Once plasma parameter estimates were finalized, these were fixed and then linked to CSF concentrations via a hypothetical effect compartment with a unidirectional rate of the entry whose rate was described by KPC and an amount, expressed as PC, or a ratio between plasma concentrations and CSF concentrations. Higher values of KPC indicate faster rates of entry, and higher values of PC indicate greater proportions of linezolid entering from the blood into the CSF.
  Parameters were estimated in NONMEM v7.5 using maximum likelihood estimation (MLE) by optimizing the likelihood function based on observed data. The First Order Conditional Estimation (FOCE) method was employed, which linearizes the model around individual-specific estimates to efficiently account for both fixed effects (population-level parameters) and random effects (individual variability).
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Linezolid
Number analyzed (Participants) | 18
ratio | .5381 [.46 to .616]

6. Secondary Outcome: Proportion of Participants With Grade 3 or Higher Adverse Events (AE).
Time Frame: 4 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Proportion of Participants Who Complete LZD Treatment.
Time Frame: 4 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Modified Rankin Scale (MRS) Performance.
Description: Measures the degree of disability/dependence on a 6 point scale ranging from 0 (no symptoms) to 6 (death).
Time Frame: 4, 12 and 24 weeks
Reporting Status: Not Posted

9. Secondary Outcome: Neurocognitive Battery Performance: Wechsler Adult Intelligence Scale-III Digit Symbol (WAIS-III).
Description: The WAIS-III assesses speed of information processing. The test consists of 133 small blank squares separated into 7 rows. Each square consists a number ranging from 1-9 and a blank space below. The participant must pair each number in the square with its corresponding symbol provided in a 'key' above the test over a time limit of 90 or 120 seconds. Scores range from 1-133 where higher scores equal indicate better outcomes.
Time Frame: 12 and 24 weeks
Reporting Status: Not Posted

10. Secondary Outcome: Neurocognitive Battery Performance: Color Trails, Part 1
Description: The Color Trails, part 1 is used to assess attention and working memory. For this test 25 circles each containing a number between 1 and 25 are randomly placed on a sheet of paper. Participants draw a line between circles as quickly as possible in numerical order. Scores are presented as time to completion. Higher values indicate greater impairment.
Time Frame: 12 and 24 weeks
Reporting Status: Not Posted

11. Secondary Outcome: Neurocognitive Battery Performance: Color Trails, Part 2
Description: The Color Trails, part 2 is used to assess executive function. For this test 25 circles each containing either a number between 1 and 13 or a letter between A through L are randomly placed on a sheet of paper. Participants draw a line between circles as quickly as possible alternating between number and letter in ascending order. Scores are presented as time to completion. Higher values indicate greater impairment.
Time Frame: 12 and 24 weeks
Reporting Status: Not Posted

12. Secondary Outcome: Neurocognitive Battery Performance: Category Fluency
Description: The Category Fluency test measures executive function and semantic fluency. Participants have 1 minute to name as many categorical items as possible. Scores are presented as the total number of correct names. Lower values indicate greater impairment.
Time Frame: 12 and 24 weeks
Reporting Status: Not Posted

13. Secondary Outcome: Neurocognitive Battery Performance: Hopkins Verbal Learning Test-Revised (HVLT-R)
Description: Either the HVLT-R or WHO-UCLA AVLT will be used to assess verbal learning and memory. In the HVLT-R Participants are asked to recall a list of 12 words. It includes four subscales: total recall, delayed recall, retention score, and recognition discrimination index. The total recall score indicates the number of correctly reported words in 3 learning trials, with a subscale ranging from 0-36. The delayed recall subscale, ranging from 0-12, indicates the number of correctly reported words in the delayed recall trial. The retention score represents the score on the delayed recall test divided by the higher of the recall scores from learning trials 2 and 3, multiplied by 100. The recognition discrimination index (RDI) is calculated by subtracting the total false positives score (semantically-related plus semantically un-related) from the total true-positives score obtained in the delayed recognition test. For all subscales, higher values indicate better outcomes.
Time Frame: 12 and 24 weeks
Reporting Status: Not Posted

14. Secondary Outcome: Neurocognitive Battery Performance: World Health Organization-University of California-Los Angeles Auditory Verbal Learning Test (WHO-UCLA AVLT).
Description: Either the HVLT-R or WHO-UCLA AVLT will be used to assess verbal learning and memory. The WHO-UCLA AVLT includes a 15 word list learned over five trials (subscale from 0-75), an interference trial (subscale from 0-15), and a 20 minute delayed recall trial (subscale from 0-15). A final delayed recognition trial is performed immediately after delayed recall. The retention score represents the score on the delayed recall test divided by the higher of the recall scores from learning trials 2-5, multiplied by 100. The recognition discrimination index (RDI) is calculated by subtracting the total false positives score from the total true-positives score obtained in the delayed recognition test. For all subscales, higher values indicate better outcomes.
Time Frame: 12 and 24 weeks
Reporting Status: Not Posted

15. Secondary Outcome: Neurocognitive Battery Performance: Grooved Pegboard Bilateral
Description: The Grooved Pegboard Bilateral test evaluates fine motor ability. One hand at a time, subjects place 25 pegs as quickly as possible in a board with randomly oriented peg holes. Scores for each hand are presented as time to completion. Higher values indicate greater impairment.
Time Frame: 12 and 24 weeks
Reporting Status: Not Posted

16. Secondary Outcome: Neurocognitive Battery Performance: Finger Tapping Bilateral
Description: The Finger Tapping Bilateral test evaluates fine motor ability. One hand at a time, subjects tap a lever counter device as quickly as possible within a 10 second time interval. A total of ten trials are conducted, five trials per hand. Trial subscores are presented as the number of taps within the 10 second interval. Trial subscores for each hand are averaged for a total score. Higher values indicate better outcomes.
Time Frame: 12 and 24 weeks
Reporting Status: Not Posted

17. Secondary Outcome: Montreal Cognitive Assessment Performance (Conditional).
Description: Completed if participant is unable to undergo the full neurocognitive test battery. The Montreal Cognitive Assessment (MoCA) is a brief cognitive screening tool used to detect mild neurocognitive disability. It assesses six key areas of cognitive ability: short-term memory, visuospatial abilities, executive functions, language, orientation to time and place, and attention, concentration and working memory. The assessment has 11 scored sections, summed for a total score ranging from 0-30 points; a score of 26 or above is considered normal.
Time Frame: 12 and 24 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | High Dose RIF With LZD | Standard Dose RIF With LZD | High Dose RIF | Standard Dose RIF
All-Cause Mortality (participants affected / at risk) | 3/9 | 3/11 | 5/10 | 4/10
Serious Adverse Events (participants affected / at risk) | 5/9 | 5/11 | 6/10 | 6/10
Other Adverse Events (participants affected / at risk) | 0/9 | 4/11 | 4/10 | 3/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose RIF With LZD (N=9) | Standard Dose RIF With LZD (N=11) | High Dose RIF (N=10) | Standard Dose RIF (N=10)
Sepsis Secondary to Multiple Pressure Sores (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unrelated to Study Drug
Drug-Induced Liver Injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Related to Study Drug
Stevens-Johnson Syndrome R/O Exfoliative Dermatitis Induced by Initiation of Zidovudine (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to Study Drug
Sepsis With Chest and Urinary Tract Focus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unrelated to Study Drug
Fever With Hyponatremia and Hypokalemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Unrelated to Study Drug
Hospitalization for Dehydration (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to Study Drug
Possible Aspiration Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Unrelated to Study Drug
Sepsis With Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unrelated to Study Drug
Aspiration Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unrelated to Study Drug
Sepsis With Chest Focus Complicated with Acute Kidney Injury and Electrolyte Imbalance (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Unrelated to Study Drug
Possible Neuro-Syphilis and Severe Hyponatremia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to Study Drug
Severe Malaria with Severe Anemia and Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Unrelated to Study Drug
Severe Malaria and Severe Anemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Unrelated to Study Drug
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — Unrelated to Study Drug
Acute Kidney Injury Secondary to Sepsis with Chest Focus (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to Study Drug
Severe Sepsis Secondary to Multi-Drug Resistant Bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unrelated to Study Drug
Severe Sepsis with Skin Focus Possible Acute Pulmonary Embolus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Unrelated to Study Drug
TB Meningitis with Moderate Hyponatremia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to Study Drug
Sepsis Secondary to Infected Decubitus Ulcer and Respiratory Failure Following Aspiration Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Unrelated to Study Drug
Sepsis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Unrelated to Study Drug
Possible Hypoglycemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Unrelated to Study Drug
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose RIF With LZD (N=9) | Standard Dose RIF With LZD (N=11) | High Dose RIF (N=10) | Standard Dose RIF (N=10)
Grade 3 or 4 anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Grade 3 or 4 hyponatremia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 4 (4) | 3 (3)
Grade 3 or 4 elevated total bilirubin (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-03): https://cdn.clinicaltrials.gov/large-docs/21/NCT04021121/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-18): https://cdn.clinicaltrials.gov/large-docs/21/NCT04021121/ICF_001.pdf